CLINICAL TRIAL: NCT05430802
Title: Furmonertinib Combined With Cisplatin/Pemetrexed as Neoadjuvant Therapy in EGFR Mutated Stage IIIA-IIIB Resectable Non-small Cell Lung Cancer (FORESEE): a Prospective, Open-label, Single-arm, Phase 2 Study
Brief Title: Neoadjuvant Furmonertinib and Cisplatin/Pemetrexed as in EGFR Mutated Stage IIIA-IIIB Resectable NSCLC (FORESEE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMR-21011
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: furmonertinib; AST2818
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib plus cisplatin/pemetrexed (Experimental): furmonertinib 80mg/d for 9 weeks and cisplatin 75mg/m2 d1 iv + pemetrexed 500mg/m2 d1 iv at 21 day cycles for 3 cycles
  Interventions: Drug: Furmonertinib+cisplating/pemetrexed

INTERVENTIONS:
Drug: Furmonertinib+cisplating/pemetrexed — Furmonertinib 80mg/d for 9 weeks and cisplating75mg/m2 d1 iv + pemetrexed 500mg/m2 d1 iv in 21-day cycles for 3 cycles

SUMMARY:
In this open-label, single-arm, phase 2 study, 40 eligible patients with EGFR mutated stage IIIA-IIIB resectable NSCLC will be recruited to receive furmonertinib for 9 weeks combined with cisplatin/pemetrexed for 3 cycles (21 d/cycle) as neoadjuvant therapy before radical surgery. Radiological and pathological evaluations will be performed before and after the neoadjuvant therapy to assess the efficacy of treatment. Adverse events during neoadjuvant therapy, disease and survival status will also be collected in the study.

ELIGIBILITY:
Inclusion Criteria:

* With written informed consent before any study procedure
* Histology or cytology diagnose of non-small cell lung cancer within 60 days
* Stage IIIA/IIIB, with resectable lesion(s) by radiology
* EGFR mutation positive (exon 19 deletions or exon 21 L858R, with or without other EGFR mutations)
* Without prior anti-tumor treatment
* With at least one measurable lesions (The longest axis ≥10mm)
* ECOG performance status 0-1
* Using adequate and effective contraception, women should refrain from breastfeeding and have a negative pregnancy test prior to the first administration of the study drug if within during child-bearing age

Exclusion Criteria:

* EGFR Exon 20 insertions positive
* Mixed with small cell cancer, or other mixed types of lung cancer
* Any prior anti-tumor treatment
* Major surgery within 4 weeks before enrolment
* Women with pregnancy or breastfeeding
* Use of strong CYP3A4 inhibitors within 7 days or strong CYP3A4 inducers within 21 days before enrolment; use of traditional Chinese medicine with anti-tumor effect within 21 days before enrolment
* With history of other malignancy except for radical resected tumors without recurrence for 5 years or more
* With severe or uncontrolled systemic disease such as uncontrolled hypertention, diabetes mellitus, chronic heart failure, unstable angina, myocardial infarction within 1 year, active hemorrhage, active HBV/HCV/HIV or other infections requiring infusion treatment
* Severe gastrointestinal diseases which may affect the intake and absorption of study drug
* Prolongation of ECG QTc or with relative risk factors
* History of interstitial lung disease or with relative risk factors
* Inadequate organ function of hematology, liver and kidney
* Allergic to study drugs or any component
* Poor adherence or other situation judged by investigator
* Patients who had participated other clinical studies of tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Approximately 9 weeks following the first dose of study drug
  The proportion of patients with complete response or partial response

SECONDARY OUTCOMES:
Major pathological response rate | Approximately 12 weeks following the first dose of study drug
  The proportion of patients with pathological response in the resected tumor
Pathological complete response rate | Approximately 12 weeks following the first dose of study drug
  The proportion of patients with pathological response rate in the resected tumor
R0 resection rate | Approximately 12 weeks following the first dose of study drugs
  The proportion of patients with R0 resection
Disease free survival | Approximately 3 years following the first dose of study drugs
  The time from enrolment to disease recurrence or death, which ever comes first
Overall survival | Approximately 5 years following the first dose of study drugs
  The time from enrolment to death of any reason
Pathological downstaging of lymph node rate | Approximately 12 weeks following the first dose of study drugs
  The proportion of patients with pathological downstaging of lymph node rate

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No